CLINICAL TRIAL: NCT04384536
Title: Effectiveness of Neural Therapy in Patients With De Quervain Tenosynovitis
Brief Title: Evaluation of Effectiveness of Local Anesthetic Injection in Patients With De Quervain Tenosynovitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hüma Bölük Şenlikci (Other)
Responsible Party: Sponsor-Investigator, Hüma Bölük Şenlikci, Principle Investigator, Baskent University Ankara Hospital
Organization: Baskent University Ankara Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26379996/79
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: De Quervain Disease
Keywords: De Quervain tenosynovitis; Local anesthetics; neural therapy
MeSH Terms: conditions — De Quervain Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural therapy group (Experimental): Neural therapy group underwent local anesthetics injections by the same physician. Local injections, segmental injections and injection of trigger points of the forearm are done. The patients are evaluated at the beginning of the study and after 4 weeks of follow-up. Pre and post-treatment visual analog scale and Duruöz Hand Index scores are obtained.
  Interventions: Procedure: Neural therapy application
- Control group (No Intervention): Control group used thumb spica splint and had rest

INTERVENTIONS:
Procedure: Neural therapy application — Local injections, C5-T8 segmental injections, trigger point injections of the forearm muscles and stellate ganglion injections are applied in each session, using a 27-gauge, 4-6 cm needle. The local injection is applied first in the first extensor compartment at the point of maximal tenderness and is directed proximally toward the radial styloid.trigger point is detected, approximately 5 mL lidocaine was injected to that point. C5-T8 segmental injections are applied intradermally to each spinous process and to 0.5-2 cm lateral of each process on the affected side. Finally, the stellate ganglion injection is applied using Fischer's modified technique.
  Arms: Neural therapy group

SUMMARY:
De Quervain tenosynovitis is the most common cause of lateral wrist pain. It occurs with stenosis of the abductor pollicis longus and extensor pollicis brevis tendons in the first dorsal extensor compartment of wrist. When these muscles are contracted, thumb extension is observed, so repeated ulnar deviation and thumb extension exacerbates pain. It is seen more commonly in middle-aged females and in the dominant hand.

Although it has been shown that fibrous tissue deposits cause thickening of the tendon sheaths, the etiology of de Quervain tenosynovitis is unclear. The prevalence of de Quervain tenosynovitis has been reported to be 0.5% in males and 1.3% in females.

Diagnosis of de Quervain tenosynovitis is based on clinical examination. The Finkelstein test is the provocation of pain with wrist ulnar deviation. Plain radiography may be useful for differential diagnosis. Conservative treatment of rest, non-steroidal anti-inflammatory drugs (NSAID), and physical therapy is applied first, then there may be a need for corticosteroid injections, and in resistant cases, surgery.

Neural therapy (NT) is a type of regulatory therapy using local anesthesia for the management of chronic musculoskeletal pain. NT includes local therapy (eg,infiltration of trigger points) and segmental therapy (eg, sympathetic ganglia, nerve roots, and peripheral nerves) . To the best of our knowledge, the effect of neural therapy on patients with De Quervain tenosynovitis has not been previously evaluated. Therefore, the aim of this study was to highlight the effect of neural therapy on this condition.

DETAILED DESCRIPTION:
In each session, 20 ml of local anesthetic (1:100 mixture of 10 mg/mL procaine) was used. Local injections, C5-T8 segmental injections, trigger point injections of the forearm muscles and stellate ganglion injections were applied in each session, using a 27-gauge, 4-6 cm needle. The local injection was applied first in the first extensor compartment at the point of maximal tenderness and was directed proximally toward the radial styloid (3 mL of the mixture). Then the forearm muscles were investigated by palpation to determine the trigger points. If any trigger point was detected, approximately 5 mL lidocaine was injected to that point. C5-T8 segmental injections were applied intradermally to each spinous process and to 0.5-2 cm lateral of each process on the affected side (approximately 0.25-0.5 ml per injection). Finally, the stellate ganglion injection was applied using Fischer's modified technique. The sternocleidomastoid muscle was palpated by the physician between the middle and distal third, gently pulling the muscle laterally with the neurovascular bundle. Following palpation of the anterior tubercle of the transverse process of the sixth cervical vertebra, the cervical spine was extended and rotated 45° to the opposite side. The needle entry point was 1 mm below the tubercle, then the needle was directed 45° caudally, 45° medially and 45° dorsally. If the aspiration was negative, 3mL procaine was injected

ELIGIBILITY:
Inclusion Criteria:

* The patients are diagnosed clinically using the Finkelstein test (in which the patient flexes the thumb and wraps the fingers over thumb, then the physician stabilizes the forearm and ulnarly deviates the wrist)
* The presence of pain over the abductor pollicis longus and extensor pollicis brevis tendons is accepted as positivity
* Patients between 18-65 years and presence of positive Finkelstein test are included the study.

Exclusion Criteria:

- Patients are excluded from the study if they have chronic widespread or local musculoskeletal pain due to rheumatological (i.e., fibromyalgia, rheumatoid arthritis), neurological diseases (i.e., multiple sclerosis, cervical discopathy or plexopathy), trauma or surgery to the related region (wrist, elbow or hand), or are aged <18 years or >65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | a month follow-up
  A 10-cm VAS was used by patients for the self-assessment of pain intensity associated with tenosynovitis. Patients were asked to score the level of pain severity on a scale marked from 0-10 where 0= no pain and 10= intolerable pain
Duruöz Hand index (DHI) | a month follow-up
  The DHI is a self-reporting scale for the evaluation of hand functions, which was first developed in 1996 for patients with rheumatoid arthritis. It consists of 18 items in 5 domains of kitchen tasks, personal hygiene, dressing, office tasks and others. Each item is scored between 0-5, to give a total score of 0-90, with higher scores indicating increased hand disability

CONTACTS AND LOCATIONS:
Overall Officials: Hüma Bölük-Şenlikci, MD, Study Director — Başkent University Medical School Hospital
Locations (1):
- Başkent University Ankara Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Before publication it would not be appropriate to share data with other researchers

REFERENCES:
- [Background] Ippolito JA, Hauser S, Patel J, Vosbikian M, Ahmed I. Nonsurgical Treatment of De Quervain Tenosynovitis: A Prospective Randomized Trial. Hand (N Y). 2020 Mar;15(2):215-219. doi: 10.1177/1558944718791187. Epub 2018 Jul 30. PMID 30060681
- [Background] Pensak MJ, Bayron J, Wolf JM. Current treatment of de Quervain tendinopathy. J Hand Surg Am. 2013 Nov;38(11):2247-9; quiz 2250. doi: 10.1016/j.jhsa.2013.06.003. Epub 2013 Jul 24. No abstract available. PMID 23890846
- [Background] Kuo YL, Hsu CC, Kuo LC, Wu PT, Shao CJ, Wu KC, Wu TT, Jou IM. Inflammation is present in de Quervain Disease--correlation study between biochemical and histopathological evaluation. Ann Plast Surg. 2015 May;74 Suppl 2:S146-51. doi: 10.1097/SAP.0000000000000459. PMID 25650747
- [Result] Egli S, Pfister M, Ludin SM, Puente de la Vega K, Busato A, Fischer L. Long-term results of therapeutic local anesthesia (neural therapy) in 280 referred refractory chronic pain patients. BMC Complement Altern Med. 2015 Jun 27;15:200. doi: 10.1186/s12906-015-0735-z. PMID 26115657